| 1 | |
|---|---|
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| 7 | |
| 8 | |
| 9 | |
| 10 | |
| 11 | A Multicenter, Partially-Masked, Randomized, Controlled Study of Medical Therapy vs. |
| 12 | Medical Therapy plus Optic Nerve Sheath Fenestration vs. Medical Therapy plus |
| 13 | Stereotactic Ventriculoperitoneal Cerebrospinal Fluid Shunting in Subjects with Idiopathic |
| 13<br>14 | Intracranial Hypertension and Moderate to Severe Visual Loss |
| 15 | |
| 16 | Surgical Idiopathic Intracranial Hypertension Treatment Trial ("SIGHT") |
| 17 | |
| 18 | STATISTICAL ANALYSIS PLAN |
| 19 | |
| 20 | Version 1.0 |
| 21 | Protocol Version 3.2 |
| 22 | |
| 23 | January 30, 2019 |
| 24 | |

# **Revision History**

The following table outlines changes made to the Statistical Analysis Plan.

| Version<br>Number | Protocol<br>Version | Author | Approver | Effective<br>Date | Study Stage | Revision Description |
|---|---|---|---|---|---|---|
| 1.0 | 3.2 | Nicole | Mike | 03-04- | No analyses | Original Version |
| 1.0 | 3.2 | Foster | McDermott | 2019 | done | Oliginal Version |

| 25 | |
|----|-------------|
| 26 | |
| 27 | |
| 28 | |
| 29 | Author: |
| 30 | |
| 31 | |
| 32 | |
| 33 | Approver: |
| 34 | |
| 35 | |
| 36 | |
| 37 | Study Lead: |
| 38 | |

## **List of Abbreviations**

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| CBC | Complete Blood Count |
| CSF | Cerebrospinal Fluid |
| D | Diopter |
| dB | Decibel |
| DSMC | Data and Safety Monitoring Committee |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| GCL | Ganglion Cell Layer |
| GEE | Generalized Estimating Equations |
| HIT-6 | Headache Impact Test |
| IIH | Idiopathic Intracranial Hypertension |
| ITT | Intention to Treat |
| MAR | Missing at Random |
| MCS | Mental Component Summary |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mm Hg | Millimeters of Mercury |
| NEI | National Eye Institute |
| ONSF | Optic Nerve Sheath Fenestration |
| PCS | Physical Component Summary |
| PMD | Perimetric Mean Deviation |
| PRC | Photography Reading Center |
| RNFL | Retinal Nerve Fiber Layer |
| SF-36v2 | Short Form Health Survey |
| VFQ-25 | Visual Function Questionnaire |
| VFRC | Visual Field Reading Center |
| VPS | Sterotactic Ventriculo-Peritoneal CSF Shunting |

#### 41 1.0 Study Overview 42 The study is a randomized trial of adults (18-<64 years old) with idiopathic intracranial 43 hypertension and moderate to severe visual loss without substantial recent treatment who are 44 randomly assigned to (1) medical therapy, (2) medical therapy plus Optic Nerve Sheath 45 Fenestration (ONSF), or (3) medical therapy plus Sterotactic Ventriculo-Peritoneal CSF 46 Shunting (VPS). 47 48 The primary study objective is to determine whether the efficacy of VPS with medical therapy is 49 superior to medical therapy alone or ONSF with medical therapy in reducing or reversing visual 50 loss in subjects with idiopathic intracranial hypertension and moderate to severe visual loss. A 51 secondary objective is to compare the treatment groups with respect to the time from 52 randomization to treatment failure over up to 3 years. 53 54 The study protocol consists of: 55 Randomized Trial 56 Screening visit 57 Baseline visit 58 Randomization 59 Safety Visits (timing dependent on treatment group) 60 • Visit 1 (4 weeks from randomization) • Visit 2 (8 weeks from randomization) 61 62 o Phone call 1 (12 weeks from randomization) 63 • Visit 3 (16 weeks from randomization) 64 o Phone call 2 (20 weeks from randomization) • Visit 4 (Primary Outcome; 26 weeks from randomization) 65 • Treatment Failure Identification Phase 66 67 o Phone call (39 weeks from randomization) • Visit 5 (52 weeks from randomization) 68 • Visit 6 (104 weeks from randomization)

71 Unscheduled visits may occur if early termination of treatment is necessary (testing will be the 72 same as the primary outcome visit).

• Visit 7 (Final visit; 156 weeks from randomization).

73 74 This document describes the analyses that will be performed.

#### 76 2.0 Sample Size

69

70

- 77 In this clinical trial, 180 subjects with newly diagnosed IIH and moderate to severe visual loss (-
- 78  $27 \text{ dB} \leq \text{PMD} \leq -6 \text{ dB}$ ) will be randomly assigned to receive either medical therapy, ONSF +
- 79 medical therapy, or VPS + medical therapy (60 per group). This sample size should provide high
- 80 power (~90%) to detect a difference in mean change of visual field between groups when the

true differences between any 2 of 3 groups is 4.5 dB with a two-tailed Bonferroni-adjusted significance level of 1.7%, allowing for an anticipated 10% drop-out. The rationale for the choice of a clinically significant treatment group difference of 4.5 dB is explained in the last paragraph of section 2.0.

The primary outcome variable in this trial will be the change from baseline to the first of Month 6 or time of treatment failure in PMD in an eligible eye. The sample size considerations initially focus on data from the best eligible eye, since most subjects are expected to contribute only one eye to the primary analysis, but addition of the other eligible eye is also considered below. In 2012, the IIH Study Group performed a retrospective chart review of consecutive newly diagnosed patients that met the modified Dandy criteria for IIH at 30 of the 41 participating sites. Data on PMD were available from 91 patients at two time points, before and after intervention, with the median follow-up time being 6.0 months (interquartile range 4.1 to 7.0 months). Patients received either medical treatment (n = 43), ONSF (n = 24), or VPS (n = 24). The mean ( $\pm$  standard deviation) changes in PMD (in dB) in the best eligible eye over the follow-up period were  $5.5 \pm 6.9$  in the medical group,  $2.0 \pm 8.9$  in the ONSF group, and  $8.2 \pm 8.0$  in the VPS group; overall these values were  $5.3 \pm 8.0$ . The distribution of these changes was slightly more peaked than would be expected for a normal distribution, as illustrated in Figure 1a and 1b.



Figure 1a and 1b. Distribution of Changes in PMD in the Best Eligible Eve

The figure on the left (a) shows the distribution of changes in PMD in the best eligible eye according to baseline PMD and intervention. Most of the patients demonstrated improvement in PMD. The figure on the right (b) shows a histogram of the changes in PMD in the best eligible eye regardless of intervention. The distribution appears to be characterized by a high concentration of changes between 0 and 10 PMD and is more peaked than normal.

Given the cross-sectional nature of the preliminary data, sample size determination based on the use of GEE for the primary analysis is very similar to that based on the use of an analysis of covariance model. If an analysis of covariance model is fit to the preliminary data, with change in PMD as the outcome variable and treatment group and baseline PMD as the independent variables, the standard deviation of the residuals is 6.3 dB. The differences between treatment groups in adjusted mean response are quite small in this analysis: -0.09 dB difference between

- the ONSF and medical groups, and 1.13 dB difference between the VPS and medical groups.
- Also, a GEE analysis produces identical adjusted group means and slightly different estimated
- standard errors than those from the analysis of covariance model.
- 114 It may be noted that the standard deviation of the residuals in the above analysis of covariance
- model is substantially less than the standard deviations in the individual treatment groups,
- reflecting adjustment for the baseline value of PMD in the analysis of covariance model and the
- fairly strong correlation between the baseline and final PMD values (r = 0.52). When considering
- only subjects who were followed for at least 5.5 months (n = 56), the correlation between the
- baseline and final PMD values was actually somewhat higher (r = 0.62) and the residual standard
- deviation in the analysis of covariance model was smaller (6.0 dB).
- 121 Assuming a standard deviation of 6.5 dB, and a Bonferroni-adjusted two-tailed significance level
- of 1.7%, in order to detect a group difference assuming a true difference of 4.5 dB with 88%
- power, a sample size of 54 subjects per group is required. The sample size will be inflated to 60
- subjects per group (180 total) to accommodate an anticipated 10% rate of subject
- withdrawal/dropout.
- The assumed standard deviation of 6.5 dB was selected based on the calculated standard
- deviation of the residuals from the above analysis of covariance model (6.3 dB) under the
- following assumptions: 1) the distribution of baseline PMD in the study cohort will be similar to
- that observed in the pilot study, and 2) the higher standard deviation observed in the pilot study
- surgical groups can be attributed to the increased probability of those with worse PMD at
- baseline to receive surgery (participants with worse PMD at baseline had higher variability of
- 132 change in PMD)<sup>a</sup>. The power remains above 80% even if the assumed standard deviation is as
- 133 large as 7.1 dB.
- The inclusion of the worst eligible eye is expected to increase power, but the increase is expected
- to be small (approximately 3%) because the preliminary data from the chart review indicate that
- only ~40% of subjects will contribute a second eligible eye to the analysis and the correlation
- between the outcomes in the two eyes is quite high (0.82 in our sample). This assumes that the
- group difference will be comparable in the best and worst eligible eyes, as we anticipate.
- The chosen effect size of 4.5 dB is based on the following rationale. Visual field defects are
- similar in IIH and glaucoma and data on the relationship between vision-specific quality of life
- 141 (as measured by the NEI-VFQ-25) and PMD from the better seeing eye are available from 213
- subjects with glaucoma in the Los Angeles Latino Eye Study. A regression analysis yielded the
- 143 finding that a change of 1 dB in PMD corresponded to an approximately one-unit score change
- on the NEI-VFO-25 composite score. In another study, Suner et al. used data from two clinical
- trials in neovascular age-related macular degeneration and anchor-based methods to estimate the
- change in NEI-VFQ-25 composite score that corresponds to a change of  $\geq$  15 letters ( $\sim$  3 lines) in
- visual acuity, a value generally accepted as clinically significant. They concluded that a change
- of 4-6 points on the NEI-VFQ-25 composite score should be considered clinically significant.
- Taken together, the results of these two investigations suggest that a change in PMD of 4.5 dB

150 corresponds to a change in NEI-VFQ-25 score that would be considered to be of minimal clinical significance. 151 152 153 <sup>a</sup>The DSMC calculated an estimated standard deviation of change in PMD of 6.9 dB based on the assumption that 154 the standard deviations in the pilot data were larger for participants who received surgery, and that the increased 155 variability was due to the surgical intervention itself. Since the surgical groups were under-represented in the pilot 156 data, the estimated variances in these groups were appropriately up-weighted in the calculation of the pooled 157 standard deviation, resulting in the estimate of 6.9 dB. The assumptions underlying the original calculation (6.5 dB) 158 and the DSMC calculation (6.9 dB) are both plausible. The DSMC agreed to move forward with the 6.5 dB standard

159

160

deviation.

#### 161 3.0 Analysis 162 163 3.1 Intention-to-Treat Principle 164 The primary statistical analyses for this trial will be performed according to the intention-to-treat 165 principle and will include all randomized subjects and eligible eyes. An eye is defined as 166 eligible if the following hold at the baseline visit: 167 Inclusion criteria 168 o Visual field loss meeting the following based on two full threshold 24-2 size V 169 tests reviewed by the Visual Field Reading Center (VFRC) 170 PMD from -6 dB to -27 dB 171 Reproducible visual loss present on automated perimetry including no 172 more than 15% false positives 173 • Visual acuity better than 20/200 (39 or more letters correct) • Exclusion criteria 174 175 o Intraocular pressure currently >28 mm Hg or >30 mm Hg at any time in the past 176 o Refractive error of more than -6.00 or more than +6.00 sphere or more than 3.00 cylinder with the following exceptions: 177 178 Eyes with more than 6.00D of myopia but less than 8.00D of myopia are eligible if: 179 180 There are no abnormalities on ophthalmoscopy or fundus photos related to myopia that are associated with visual loss (such as 181 182 staphyloma, retinal thinning in the posterior pole, or more than mild optic disc tilt), and 183 • The individual will wear a contact lens for all perimetry 184 185 examinations with the appropriate correction Eyes with more than 6.00D of hyperopia but less than 8.00D of hyperopia 186 are eligible if: 187 188 • There is an unambiguous characteristic halo of peripapillary edema 189 as opposed to features of a small crowded disc or other hyperopic 190 change related to visual loss determined by the Site Investigator or 191 the PRC Director (or his designate), and • The individual will wear a contact lens for all perimetry 192 193 examinations with the appropriate correction (which can be 194 corrected for perimetry or the patient's own contact lens with over 195 correction by lens at perimeter) o Other disorders causing visual loss except for refractive error and amblyopia, 196 197 including cells in the vitreous or iritis

o Large optic disc drusen on exam or in previous history (small drusen of the disc

investigator determines they are contributing to vision loss).

can occur with longstanding papilledema and are allowed if not so numerous that

198

199

Every effort will be made to retain subjects in this study, to promote adherence to the study protocol, and to collect all data at every visit. If a subject cannot tolerate study medication or refuses to receive the study intervention, we will continue to follow and evaluate that subject if he/she is willing. If a subject drops out, attempts will be made to bring the subject back for a final evaluation. Compliance with trial procedures, drop-outs/drop-ins, and reasons for subject withdrawal will be carefully tracked throughout the study.

#### 3.2 Analysis of the Primary Outcome Variable

#### 3.2.1 Definition of Primary Outcome

The primary outcome variable will be the change from baseline to first of Month 6 or time of treatment failure in PMD in an eligible eye, with data from all eligible eyes included in the primary analysis (refer to the table below for a description of eyes included in the primary analysis).

| Eyes at baseline | Eyes included in primary analysis |
|---|---|
| No eligible eyes → subject not eligible | None (subject not eligible) |
| One eligible eye and non-eligible eye too good | One eye that was eligible at baseline, regardless of what happened to either eye during study |
| One eligible eye and non-eligible eye too bad | One eye that was eligible at baseline, regardless of what happened to either eye during study |
| Two eligible eyes | Both eyes that were eligible at baseline, regardless of what happened to either eye during study |

Treatment of subjects who have reached criteria for treatment failure will be at the discretion of the Site Investigator, and this treatment may yield a different outcome than randomized treatment. For this reason, the primary outcome variable for subjects who reach criteria for treatment failure prior to Month 6 will be the PMD measured at the time of treatment failure for purposes of the primary analysis. It is anticipated that no more than 15% of subjects will reach criteria for treatment failure prior to Month 6.

- 225 PMD (baseline or outcome) will be the average PMD from the two reliable visual field
- examinations (i.e. meeting Visual Field Reading Center criteria) performed at the visit; if only
- one reliable result is obtained on the visual field examination, the one reliable result will be
- analyzed; if a reliable result is not obtained on the visual field examinations, the PMD will be
- 229 considered missing.

- Outcome PMD (excluding PMD at time of treatment failure) from visual field testing performed
- out of the window of 168-242 days from randomization will be considered missing for the
- primary analysis. Note this means a subject can be up to two weeks early and up to a full 60
- days late, this latter choice was made with clinician input that they would rather have a
- 235 measurement than impute.

236237

#### 3.2.2 Primary Statistical Model

- The primary statistical analysis will involve fitting an analysis of covariance model using
- 239 generalized estimating equations (GEE) with treatment group as the factor of interest and
- baseline PMD as a covariate. These analyses will accommodate correlation among the within-
- subject responses between the two eyes; an exchangeable working correlation structure will be
- used. Standard errors for the model parameters will be estimated using the robust "sandwich"
- estimators. The model also does not rely on the assumption of normality.
- 244 This model will be used to determine Bonferroni-adjusted confidence intervals for the three pair-
- 245 wise differences among the adjusted treatment group mean responses (treatment effects);
- likewise, tests will be performed to compare the adjusted treatment group means using a
- Bonferroni-adjusted two-tailed significance level. An overall confidence coefficient of 98.3%
- and corresponding significance level of 1.7% for each comparison will be maintained, but as
- 249 discussed in section 3.7.2 below, the confidence coefficient for interval estimation and
- significance level for hypothesis testing will be adjusted for the interim analysis for efficacy.

251252

#### 3.2.3 Adjustment for Baseline Characteristics

- 253 Baseline characteristics of subjects will be summarized overall and by treatment group. Formal
- statistical comparisons between treatment groups will not be performed; instead, potential
- 255 confounding will be explored by examination of the magnitudes of treatment group differences
- in the distributions of visual acuity, papilledema grade, and duration of IIH. Other variables for
- 257 which there are baseline differences among treatment groups that could be associated with the
- outcome also will be evaluated for a potential confounding effect. Continuous variables will be
- described using means, standard deviations, medians, quartiles, and ranges, and categorical
- variables will be described using percentages.
- 261 If clinically important differences are found between the groups at baseline, the primary outcome
- analyses will be repeated after statistically adjusting for these differences. These analyses will be
- 263 considered secondary, however.

### 3.2.4 Investigation of Treatment by Covariate Interactions

- We will investigate the interaction between treatment group and selected baseline covariates
- 267 (age, race/ethnicity, PMD (average of measures from two reliable visual field examinations),
- 268 papilledema grade, RNFL thickness, total retinal thickness, optic nerve head volume, visual
- acuity, presence of transient visual obscurations, and the symptom of constant visual loss)
- separately by adding the appropriate main effect and interaction terms to the primary statistical
- 271 model and testing for significance of the interaction.
- 272 Since the power to detect potentially meaningful interactions will be limited, the magnitudes of
- 273 mean responses to treatment in the relevant subgroups will be examined. The observation of
- 274 clinically important subgroup differences in mean treatment response will serve as hypothesis
- 275 generation for possible future studies designed to address specifically the issue of differential
- therapeutic response. Although these analyses are purely exploratory, those involving
- papilledema grade, PMD, visual acuity, and race/ethnicity will be given higher priority.
- 278 Interpretation of subgroup analyses should be viewed with caution, irrespective of whether the
- overall analysis demonstrates a significant treatment group difference. Extreme caution is
- particularly needed in the absence of such an overall difference.

281282

#### 3.2.5 Verification of Model Assumptions

- The underlying assumptions of the statistical model to be used in the primary analysis will be
- 284 thoroughly checked (e.g., linearity) through assessment of scatterplots of change in PMD versus
- baseline PMD within treatment group, and remedial measures (e.g., inclusion of baseline PMD
- 286 categorized according to randomization strata) may be taken if serious violations of these
- assumptions are detected.

288289

#### 3.2.6 Treatment of Missing Data

- 290 Multiple imputation will be used to deal with missing data. This will be applied using a
- regression-based imputation model. For subjects with complete data up to a particular visit, a
- linear regression model (identity link) will be fit that includes the outcome at that visit as the
- 293 dependent variable and outcomes at previous visits and treatment group as independent
- variables. Separate models will be similarly constructed for each visit (Weeks 4, 8, 16, and 26).
- Using these regression models, a missing value for a subject at a particular visit will be imputed
- as a draw from the predictive distribution given the outcomes at previous visits (some possibly
- imputed) and treatment group. This will be done sequentially starting with the Week 4 visit and
- ending with the Week 26 (Month 6) visit. This process will be repeated 100 times, resulting in
- 299 100 complete analysis data sets. The analyses (Section 3.2.2) will be performed separately for
- 100 complete analysis data sets. The analyses (Section 3.2.2) will be performed separately for
- and the results will be combined into one multiple
- imputation inference (estimated treatment effect and associated confidence interval and p-value)
- 302 using Rubin's rules. This approach is appropriate for data sets that have a monotone missing

data pattern. If the data set does not precisely have this pattern, the monotone data augmentation method using Markov-Chain Monte-Carlo as proposed by Li (1988) and Liu (1993) will be used to impute the small amount of missing data that is required to make the missing data pattern monotone before applying the multiple imputation algorithm described above. This approach should accommodate missing data in an appropriate way under the missing at random (MAR) assumption.

309310

311

312

313

314

315

316

317

318

319

320

321

322

323

#### 3.2.7 Sensitivity Analysis

- The primary analysis will be completed using the ITT principle described in *Section 3.1*. The primary analysis will be repeated with the following considerations as a secondary analysis:
  - According to treatment received (whether or not this was the randomly assigned treatment)
    - Excluding participants without outcome PMD (Month 6 or exam at early treatment failure)
    - Exclude participants who took less than 80% of tolerated dosage of medication
    - Exclude participants with major protocol violations such as: receipt of additional treatment outside of treatment assignment prior to first of 6-month visit or visit at which treatment failure declared, or major eligibility deviation that could impact the ability to assess the primary outcome.
  - The identification of subjects to be excluded from these analyses will be determined before the masking is broken (i.e., before data analysis).

324

# 325326

327

328

329

330

331

332

333

334

335

336

337

338

339

340

341

#### 3.3 Analysis of Secondary Outcome Variables for Efficacy

#### 3.3.1 Definition of Secondary Outcomes

- The following are secondary outcomes for efficacy:
  - Change from baseline PMD to Month 6 PMD
    - o PMD defined as described in Section 3.2.1
    - Month 6 PMD value will be used even for participants with treatment failure prior to Month 6
  - Change from baseline to Month 6 CSF opening pressure measurement by lumbar puncture
  - Change from baseline to Month 6 in papilledema grade
    - Papilledema grade determined by reading center and grade determined by study center will be considered separate outcomes and will be analyzed separately
  - Change from baseline to Month 6 (pre-lumbar puncture) in RNFL thickness
  - Change from baseline to Month 6 (pre-lumbar puncture) in total retinal thickness
  - Change from baseline to Month 6 (pre-lumbar puncture) in optic nerve head volume
  - Change from baseline to Month 6 (pre-lumbar puncture) in ganglion cell layer thickness

342 • Change from baseline to Month 6 (pre-lumbar puncture) in optic nerve canal shape • Change from baseline to Month 6 in ETDRS visual acuity score 343 344 • Change from baseline to Month 6 in SF-36v2 scores 345 o Change will be calculated separately for each of the eight health domains and the 346 physical component summary (PCS) and mental component summary (MCS) 347 scores 348 Scores determined via SF-36v2 scoring software 349 Change from baseline to Month 6 in VFQ-25 score 350 Score determined as an average of sub-scale scores as described in the VFQ-25 351 manual (..\..\References\Participant Questionnaires\VFQ25 Manual.pdf) 352 Scoring of missing items will follow the scoring instrument 353 Change from baseline to Month 6 in VFQ-25 Neuro-Ophthalmic Supplement score 354 o Score determined as described in the 10-item Neuro-Ophthalmic instructions 355 (..\.\References\Participant Questionnaires\Prior to Executed 356 Agreement\10ItemNeuroOpthalVFQ25.pdf) 357 Scoring of missing items will follow the scoring instrument 358 Change from baseline to Month 6 in HIT-6 Score determined as a sum of scores for each question (Never = 6, Rarely = 8, 359 Sometimes = 10, Very Often = 11, Always = 13; total score range 36 to 78 with 360 higher score indicating greater life impact) 361 362 o Surveys with >1 missing responses will be given an overall null score for the visit • Change in headache severity from baseline to Month 6 as reported on the Headache 363 364 Assessment form 365 o Analyzed as a continuous value with the following categories assigned for 366 display: 367 Mild = score 1-4 | Moderate = score 5-7 | Severe = score 8-10 368 • Month 6 VFRC determination of whether the visual field examination has improved, 369 remained the same, or worsened 370 o All available visual field examinations will be analyzed. For the initial secondary

outcome, the Month 6 VFRC rating will be used; a supplemental secondary

outcome will use the VFRC rating at time of treatment failure for subjects

experiencing treatment failure prior to Month 6.

Change in weight from baseline to Month 6

- 371
- 372373
- 374
- 375 376
- Data from all eligible eyes will be included in the analysis. With the exception of CSF opening pressure and VFRC determination of visual field status, the outcomes also will be examined with
- 377 378
- 379380
- 3.3.2 Secondary Statistical Models

change from baseline to Months 12, 24, 36.

- 381 Treatment effect on secondary outcome variables for efficacy that are continuous will be
- analyzed using the same methods described in Section 3.2.2 for the primary outcome variable,
- except that a working correlation structure will not be needed for variables that are not eye-
- specific. Variables to be analyzed in this manner are:
- Change in PMD at Month 6
  - Change in CSF opening pressure (does not require working correlation structure)
- Change in papilledema grade (both reading center and study center outcomes)
- Change in RNFL thickness
  - Change in total retinal thickness
    - Change in optic nerve head volume
- Change in ganglion cell layer thickness
- Change in optic nerve canal shape
  - Change in ETDRS visual acuity score
  - Change in SF-36 scores (8 subscale domains, PCS and MCS; does not require working correlation structure)
    - Change in VFQ-25 score (does not require working correlation structure)
    - Change in VFQ-25 Neuro-Ophthalmic Supplement score (does not require working correlation structure)
  - Change in HIT-6 (does not require working correlation structure)
    - Change in headache severity as reported on Headache Assessment form (does not require working correlation structure)
      - Change in weight

405

406

407

386

389

390

393

394

395

396

397

398

399

400

401

402

The treatment effect on the ordinal outcome of Month 6 visual field examination status by the VFRC (improved, no change, worse) will be assessed via a logistic regression model (proportional odds model). A likelihood ratio test will be performed for significance of the adjusted treatment group odds ratios representing pair-wise treatment group comparisons; 98.3% confidence intervals will be constructed for these odds ratios.

408 409 410

411

412

All models will include treatment group as the factor of interest and the baseline value of the outcome variable as a covariate (to replace baseline PMD adjustment in the primary for continuous outcomes; Month 6 visual field examination status by VFRC will retain inclusion of baseline PMD).

413 414 415

#### 3.3.3 Adjustment for Baseline Covariates

Assessment for and implementation of adjustment for baseline covariates will follow methods described in *Section 3.2.3*.

418 419

#### 3.3.4 Investigation of Treatment by Covariate Interactions

| 420<br>421<br>422 | methods described in <i>Section 3.2.4</i> . |
|---|---|
| 423 | 3.3.5 Verification of Model Assumptions |
| 424 | Methods described in <i>Section 3.2.5</i> will be used to check underlying assumptions of the |
| 425 | statistical model for each outcome. |
| 426 | |
| 427 | 3.3.6 Treatment of Missing Data |
| 428 | Methods described in Section 3.2.6 will be used to impute missing data at Month 6 for |
| 429 | continuous outcomes. |
| 430 | |
| 431 | Missing values of Month 6 visual field examination status will not be imputed. |
| 432 | |
| 433 | 3.4 Compliance Outcomes |
| 434 | Data concerning compliance with acetazolamide (pill counts, serum bicarbonate levels) and |
| 435 | surgical therapy will be summarized by treatment group and visit. Subjects with two eligible |
| 436 | eyes will have this information summarized by eye as well as by treatment group and visit. |
| 437 | |
| 438 | 3.5 Analysis of Safety and Tolerability Outcomes |
| 439 | 3.5.1 Adverse Events |
| 440 | All reportable adverse events will be tabulated by treatment group in a listing of each reported |
| 441 | Medical Dictionary for Regulatory Activities (MedDRA) term and summarized over each |
| 442 | MedDRA System Organ Class. Details will be provided in a listing of each event. |
| 443<br>444 | In addition, the following will be tabulated by treatment group. When applicable, events will be tabulated by eye within person: |
| 445 | <ul> <li>Number of adverse events per subject</li> </ul> |
| 446 | <ul> <li>Number of subjects with at least one event</li> </ul> |
| 447 | • |
| 448 | <ul> <li>Number of subjects with at least one event per person-month (person-month based on<br/>subject duration in the study)</li> </ul> |
| 449 | <ul> <li>Number of serious adverse events per subject</li> </ul> |
| 450 | <ul> <li>Number of subjects with at least one serious adverse event</li> </ul> |
| 451<br>452 | <ul> <li>Number of hospitalizations and reasons for the hospitalization (overall and per subject,<br/>separately)</li> </ul> |
| 453<br>454 | <ul> <li>Number of adverse events thought by investigator to be related to study drug and<br/>frequency of each type of such event</li> </ul> |
| 455 | <ul> <li>Number of subjects who stopped the intervention in response to an adverse event</li> </ul> |

- 456 For binary variables (occurrence of at least one event, occurrence of at least one serious adverse
- event, occurrence of at least one hospitalization, occurrence of at least one adverse event related
- 458 to treatment, occurrence of stopping the intervention in response to adverse event), Fisher exact
- 459 tests will be used to compare treatment groups. For counts (number of adverse events per
- subject, number of serious adverse events per subject, number of hospitalizations per subject),
- 461 groups will be compared using Poisson regression with inclusion of the logarithm of study
- follow-up duration for the participant as an offset term; a negative binomial model will be
- considered if overdispersion is present, and a zero-inflated negative binomial model will be used
- if there appear to be excessive zero counts.
- For each adverse event, the treatment groups will be compared in a pair-wise fashion regarding
- the occurrence of at least one event using Fisher's exact tests; numbers of individual events will
- also be described. The comparisons will be repeated excluding all mild symptoms. Similar
- analyses will be performed after grouping adverse events by body system using Medical
- Dictionary for Regulatory Activities (MedDRA) coding. All subjects will be included in these
- analyses.

#### 3.5.2 Laboratory Test Results and Vital Signs

- 473 Continuous measures of safety such as laboratory test results (CBC with platelet count,
- electrolytes, potassium, bicarbonate, and liver function tests) and vital signs and anthropometric
- 475 measures (blood pressure, weight, and waist circumference) will be analyzed descriptively
- 476 through summary statistics and tabulations.
- 477 Proportions of subjects with particular laboratory test abnormalities will be compared between
- 478 the treatment groups in a pair-wise fashion using Fisher's exact tests.

479 480

#### 3.6 Analysis of Long-Term Follow-Up Data

- The following outcome will be examined in analysis of long-term follow-up data:
  - Time from randomization to treatment failure

482 483

484

## 3.6.1 Analysis Model

- 485 Treatment group differences with respect to long-term outcomes will be assessed by fitting a Cox
- 486 proportional hazards regression model with treatment group as the factor of interest and baseline
- PMD in the best eligible eye as a covariate. Due to the discrete time data, Efron approximation
- will be used to deal with tied event times. The model will be used to determine Bonferroni-
- adjusted 98.3% confidence intervals for the adjusted hazard ratios for the three pair-wise
- 490 treatment group comparisons. Likewise, likelihood ratio tests will be performed for the
- 491 significance of these hazard ratios using a Bonferroni-adjusted two-tailed significance level of
- 492 1.7%. Kaplan-Meier curves will be used to describe the cumulative probability of treatment
- failure over time in each treatment group.

For subjects who do not experience the outcome, event times will be censored at the last subject contact at which the subject was determined to not have experienced the outcome (e.g., at time of premature withdrawal from the trial or at the final trial visit).

498 499

500

501

502

#### 3.6.2 Adjustment for Baseline Covariates

Adjustment for additional baseline covariates (in addition to baseline PMD and papilledema grade in best eligible eye) may be considered depending on the comparability of the treatment groups at baseline (refer to *Section 3.2.3*).

503504505

506

507

#### 3.6.3 Investigation of Treatment by Covariate Interactions

Examination of interactions between treatment group and selected baseline covariates will be performed using the Cox proportional hazards model following the guidelines established in *Section 3.2.4*.

508509510

### 3.6.4 Verification of Model Assumptions

The underlying assumptions of the Cox proportional hazards model will be checked and a thorough analysis of the martingale residuals and other diagnostics will be performed. Remedial measures (covariate transformation) will be taken if serious violations of these assumptions are detected.

515

The proportional hazards assumption will be assessed graphically by plotting log( $-log(\hat{S}(t))$  vs. log(time) for each of the treatment groups, and by examining plots of smoothed Schoenfeld residuals. The assumption also will be examined by dividing the time scale into 6-month periods and estimating the treatment group hazard ratios separately in each of these periods through the use of time-dependent covariates. The period length of 6 months may be adjusted prior to unmasking, based on the observed distribution of event times, if relatively few events occur during 6-month periods. Treatment group comparisons will be described in this manner if the

523 proportional hazards assumption appears to be seriously violated.

The assumption of independence between censoring time and the (unobserved) event time will be assessed by performing a sensitivity analysis in which subjects with event times that are censored prior to their scheduled end of follow-up will be treated as having experienced the event a short time (one week) after censoring.

529530

524

#### 3.7 Interim Analysis

## **3.7.1 Interim Analysis for Safety**

Interim analyses of safety data will be performed periodically throughout the trial. While the safety of subjects will be the primary concern of the DSMC, it is difficult to formulate precise

- stopping guidelines that would cover all of the possible situations that might arise. Adverse
- events, particularly serious adverse events and surgical complications, will have to be considered
- carefully by the DSMC in terms of treatment group imbalances and severity. Events of particular
- concern include the following: death, absence of light perception, hypokalemia (from Lasix use),
- surgery-associated visual loss (from either VPS or ONSF), fenestration failure and orbital
- infection (from ONSF), and shunt failure, infection, seizures, and subdural hematoma (from
- 540 VPS). If potential safety concerns are identified, the DSMC may require review of visual field
- data in order to evaluate the risk-benefit of continuing the trial as planned or modifying (or
- halting) the trial.

#### 3.7.2 Interim Analysis for Efficacy

- We will perform a single interim analysis for efficacy based on the primary outcome efficacy
- variable. This will be performed after ~50% of the subjects have completed (or were scheduled
- to have completed, based on their randomization date) their Month 6 visit and will only include
- data from these subjects. Given that recruitment of the 180 subjects will take place over 3 years,
- assuming that recruitment is uniform over time, it is anticipated that slightly fewer than 70% of
- the subjects will be enrolled at the time of the interim analysis.
- The analysis will involve pair-wise comparisons among the treatment groups with respect to the
- primary outcome efficacy variable; the significance level used for each comparison will be
- 553 determined by an O'Brien-Fleming α-spending function for a two-group comparison divided by
- 3 (Bonferroni correction). In this case, the boundaries will be Z = 3.394 for the interim analysis
- and Z = 2.400 for the final analysis. Assuming that there are 30 subjects per group and that the
- standard deviation is 6.5 dB at the interim analysis, the boundary will be crossed if a group
- difference exceeds approximately 5.7 dB. This monitoring procedure will have a negligible
- impact on the overall Type I error probability: the significance level at the final analysis
- corresponding to Z = 2.400 is  $\alpha = 0.0164$ . Point and interval estimates of treatment effects for the
- primary analysis, as well as reported p-values, will be adjusted for the interim analysis. The bias-
- adjusted mean will be used for point estimation and confidence intervals and p-values based on
- the MLE (sample mean) ordering of the sample space defined by the group sequential design
- will be reported.
- The efficacy boundary will be considered to be non-binding. We believe that it may be prudent
- to halt or modify the trial only if (1) two of the treatment groups are each shown to be superior to
- the third (in which case the third group may be dropped) or (2) one of the treatment groups is
- shown to be superior to each of the other two (in which case the trial may be halted). Of course,
- the relative safety profiles of the treatments would have to factor into these considerations as
- 569 well.

570

571572

#### 3.8 Additional Tabulations

- A flow chart will track all participants who were enrolled, indicating the reason for any who did
- not complete the study and providing details on randomized subjects determined to be ineligible.
- A summary of safety visits, phone calls, and information on completion of questionnaires will be
- 576 compiled.

579

580 581

582

- 578 Tabulations will include:
  - Demographic and clinical characteristics at enrollment by treatment group
  - Eligible eye characteristics by treatment group
    - Non-eligible eye characteristics by treatment group
    - Overall number of treatment failures by treatment group
- Overall number of surgical malfunctions by treatment group (ONSF and VPS groups)
- Duration (days) from enrollment to randomization
  - Duration (days) from randomization to surgery (ONSF and VPS groups)

585 586 587

588

589

590591

595

600

601

602 603

## **Specific Protocol Tabulations by Treatment Group**

#### 6-Month RCT

- Receipt of surgery other than that randomly assigned
- Adherence to medical management and diet by visit
- Daily dosage of acetazolamide and furosemide prescribed at each visit
- Medical therapy at each visit
- ONSF completion status (ONSF group)
- VPS completion status (VPS group)
  - Surgical complications (separately for ONSF and VPS groups)
- Reoperations (ONSF)
- Shunt revisions (VPS)
- Headache by visit
- Weight by visit
  - Visual field at follow-up (eligible eyes and non-eligible eyes, separately)
  - Visual acuity at follow-up (eligible eyes and non-eligible eyes, separately)
  - Papilledema grading at follow-up (eligible eyes and non-eligible eyes, separately)
    - RNFL and macula GCL at follow-up (eligible eyes and non-eligible eyes, separately)
  - Protocol deviations

604 605 606

607 608

#### Treatment Failure Identification Phase (Post 6-Month RCT)

- Adherence to medical management and diet by visit
- Daily dosage of acetazolamide and furosemide prescribed at each visit
- Medical therapy at each visit
- Protocol deviations.